CLINICAL TRIAL: NCT04203537
Title: A Two-Part, Phase 1/2, Randomized, Double-blind, Placebo-Controlled, Adaptive Safety, Pharmacokinetics and Preliminary Efficacy Study of CA-008 in Patients Undergoing Total Knee Arthroplasy
Brief Title: Study Evaluating the Safety, Efficacy and Pharmacokinetics of CA-008 (Vocacapsaicin)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Concentric Analgesics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA-PS-208
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Postsurgical Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Part A: dose ascending, placebo-controlled Part B: randomized, double-blind, placebo-controlled, parallel design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CA-008 36 mg (Active Comparator): Single administration (0.3 mg/mL concentration)
  Interventions: Drug: CA-008
- CA-008 60 mg (Active Comparator): Single administration (0.5 mg/mL concentration)
  Interventions: Drug: CA-008
- CA-008 90 mg (Active Comparator): Single administration (0.75 mg/mL concentration)
  Interventions: Drug: CA-008
- Placebo (Placebo Comparator): Single administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CA-008 — Local administration during surgery
  Other Names: vocacapsaicin
  Arms: CA-008 36 mg; CA-008 60 mg; CA-008 90 mg
Drug: Placebo — Local administration during surgery
  Arms: Placebo

SUMMARY:
In the pilot (Part A) of this study, multiple doses of CA-008 (vocacapsaicin) were evaluated for safety, tolerability, and PK. Doses were then selected for the expanded part (Part B) of the study, where CA-008 was compared to placebo. Patients had serial assessments of safety, PK, and drug effect.

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

* Scheduled elective Total Knee Arthroplasty (TKA) under spinal anesthesia
* Aged 18-80 years old
* ASA physical class 1, 2, or 3
* BMI </= 42 kg/m2
* Generally healthy

Exclusion Criteria:

* Concurrent condition requiring analgesic treatment during study period
* Opioid tolerant
* Known allergy to capsaicin or other study medication
* Use of prohibited medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daneshvari Solanki, MD, Principal Investigator — HD Research
Locations (4):
- United States (4):
  - Lotus Clinical Reserach, LLC, Pasadena, California
  - Legent Orthopedic Hospital, Carrollton, Texas
  - First Surgical Hospital, Houston, Texas
  - Plano Surgical Hospital, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A consisted of 3 small, sequential, placebo-controlled, dose-escalation cohorts evaluating 36, 60 and 90 mg for safety. Part B evaluated 36 and 60 mg compared to placebo in parallel, randomized groups. Efficacy data from Part A remained blinded until the end of Part B and these data were pooled for analysis.
Pre-assignment Details: Of the 193 enrolled participants, 193 met inclusion criteria and were randomized to treatment. 1 patient randomized to the 36 mg cohort and 1 patient randomized to the 60 mg cohort received placebo. These two patients were included in the placebo group. The efficacy and safety data from Parts A and B of the study are pooled by treatment group for the placebo, 30 mg and 60 mg treatment groups.
Groups:
- CA-008 36 mg (Patients From Part A); CA-008 60 mg (Patients From Part A); CA-008 90 mg (Patients From Part A); CA-008 36 mg (Patients From Part B); CA-008 60 mg (Patients From Part B): Single administration
  CA-008 (vocacapsaicin): Local administration during surgery
- Placebo (Patients From Part A); Placebo (Patients From Part B): Single administration
  Placebo: Local administration during surgery
Period: Overall Study
Arm/Group | CA-008 36 mg (Patients From Part A) | CA-008 60 mg (Patients From Part A) | CA-008 90 mg (Patients From Part A) | Placebo (Patients From Part A) | CA-008 36 mg (Patients From Part B) | CA-008 60 mg (Patients From Part B) | Placebo (Patients From Part B)
Started | 6 | 6 | 6 | 6 | 54 | 55 | 60
Completed | 6 | 6 | 6 | 6 | 54 | 55 | 60
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 subject was randomized to CA-008 60 mg, but actually received placebo
  1 subject was randomized to CA-008 36 mg, but actually received placebo
  Both subjects are included in the placebo arm
Groups:
- CA-008 36 mg; CA-008 60 mg; CA-008 90 mg: Single administration
  CA-008: Local administration during surgery
- Total: Total of all reporting groups
Arm/Group | CA-008 36 mg | CA-008 60 mg | CA-008 90 mg | Placebo | Total
Number analyzed (Participants) | 60 | 61 | 6 | 66 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (7.79) | 63.1 (7.82) | 65.5 (8.92) | 59.7 (6.45) | 62.3 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 4 | 39 | 104
  Male | 31 | 29 | 2 | 27 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 16 | 0 | 12 | 39
  Not Hispanic or Latino | 49 | 45 | 5 | 54 | 153
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 2 | 5 | 1 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 10 | 0 | 9 | 32
  White | 45 | 45 | 5 | 56 | 151
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Scores
Description: Mean area under the curve (AUC) of the Numeric Rating Scale (NRS) weighted sum of pain intensity scores (at rest) from 0-10 where 0 is no pain and 10 is the worst pain imaginable for CA-008 compared to placebo. AUC is calculated using the standard trapezoidal rule from serial measures of NRS taken every 4 hours from 0-96 hours following surgery and twice daily from 96h to Day 15
Time Frame: 0 to Day 15 post dose
Population: 193 patients - Modified Intent-to-Treat
  One patient who was randomized to CA-008 36 mg, but actually received Placebo is included in CA-008 36 mg.
  One patient who was randomized to CA-008 60 mg, but actually received Placebo is included in CA-008 60 mg.
Measure: Mean (Standard Deviation); unit: scores on a scale*hours
Groups:
- CA-008 36 mg (0.3 mg/mL Concentration); CA-008 60 mg (0.5 mg/mL Concentration); CA-008 90 mg (0.75 mg/mL Concentration): Single administration
  CA-008: Local administration during surgery
Arm/Group | CA-008 36 mg (0.3 mg/mL Concentration) | CA-008 60 mg (0.5 mg/mL Concentration) | CA-008 90 mg (0.75 mg/mL Concentration) | Placebo
Number analyzed (Participants) | 61 | 62 | 6 | 64
scores on a scale*hours
  AUC 12-96 hour | 367.41 (137.561) | 415.27 (140.967) | 373.92 (175.834) | 447.05 (108.596)
  AUC 0-96 hour | 397.68 (152.002) | 448.02 (155.948) | 403.08 (172.515) | 481.97 (120.535)
  AUC 0-Day 15 | 1235.36 (608.259) | 1530.93 (571.337) | 1629.97 (437.951) | 1452.08 (493.622)
Statistical Analysis 1: Comparison: CA-008 36 mg (0.3 mg/mL Concentration) vs Placebo; Test type: Superiority; p = 0.0004, ANOVA

2. Secondary Outcome: Total Opioid Consumption
Description: CA-008 versus placebo comparison, total opioid consumption in oral morphine equivalents
Time Frame: 0 to Day 15 post dose
Population: 193 patients - Modified Intent-to-Treat One patient who was randomized to CA-008 36 mg, but actually received Placebo is included in CA-008 36 mg. One patient who was randomized to CA-008 60 mg, but actually received Placebo is included in CA-008 60 mg.
  Opioid consumption (OC) in oral morphine equivalent dose (OME)
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Arm/Group | CA-008 36 mg (0.3 mg/mL Concentration) | CA-008 60 mg (0.5 mg/mL Concentration) | CA-008 90 mg (0.75 mg/mL Concentration) | Placebo
Number analyzed (Participants) | 61 | 62 | 6 | 64
mg morphine equivalents
  OC12-96 hours | 141.37 (75.98) | 165.92 (81.48) | 151.04 (70.59) | 206.26 (82.11)
  OC0-96 hours | 154.795 (85.95) | 183.74 (89.74) | 177.29 (66.67) | 219.94 (88.19)
  OC 0- Day 15 | 206.04 (132.99) | 275.07 (155.14) | 263.54 (138.11) | 319.12 (164.62)
Statistical Analysis 1: Comparison: CA-008 36 mg (0.3 mg/mL Concentration) vs Placebo; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: CA-008 60 mg (0.5 mg/mL Concentration) vs Placebo; Test type: Superiority; p = 0.0026, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 76 days for participants in the study. This was comprised of a screening period that could be up to 45 days and subsequent clinic visits through Day 29.
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information in this study did not differ from the clinicaltrials.gov definitions.
Arm/Group | CA-008 36 mg | CA-008 60 mg | CA-008 90 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/61 | 0/6 | 0/66
Serious Adverse Events (participants affected / at risk) | 2/60 | 1/61 | 0/6 | 2/66
Other Adverse Events (participants affected / at risk) | 54/60 | 58/61 | 6/6 | 66/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CA-008 36 mg (N=60) | CA-008 60 mg (N=61) | CA-008 90 mg (N=6) | Placebo (N=66)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CA-008 36 mg (N=60) | CA-008 60 mg (N=61) | CA-008 90 mg (N=6) | Placebo (N=66)
Bradycardia (Cardiac disorders) | 3 (3) | 4 (4) | 0 (0) | 5 (5)
Tachycardia (Cardiac disorders) | 13 (13) | 17 (17) | 3 (3) | 12 (12)
Constipation (Gastrointestinal disorders) | 29 (29) | 32 (32) | 4 (4) | 30 (30)
Nausea (Gastrointestinal disorders) | 24 (24) | 28 (28) | 5 (5) | 36 (36)
Vomiting (Gastrointestinal disorders) | 9 (9) | 11 (11) | 1 (1) | 15 (15)
Drug ineffective (General disorders) | 3 (3) | 3 (3) | 1 (1) | 7 (7)
Pyrexia (General disorders) | 12 (12) | 10 (10) | 2 (2) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 1 (1) | 5 (5)
Dizziness (Nervous system disorders) | 8 (8) | 2 (2) | 2 (2) | 7 (7)
Headache (Nervous system disorders) | 5 (5) | 7 (7) | 0 (0) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 1 (1) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 9 (9) | 2 (2) | 10 (10)
Hypertension (Vascular disorders) | 3 (3) | 5 (5) | 0 (0) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infusion site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Incision site discharge (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incision site vesicles (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural oedema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Blood pressure increased (Investigations) | 2 (2) | 3 (3) | 0 (0) | 4 (4)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diastolic hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT04203537/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT04203537/SAP_001.pdf